CLINICAL TRIAL: NCT05727085
Title: Cohort of Twin Pregnancy and the Offspring
Acronym: CTPO
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Xiong, Clinical Professor, Fudan University
Other Study IDs: TW20231535
Record Dates: First submitted 2022-10-23; First posted 2023-02-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-07

CONDITIONS: Twin Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- twins
  Interventions: Other: All pregnant women with a twin pregnancy and the offspring

INTERVENTIONS:
Other: All pregnant women with a twin pregnancy and the offspring — No intervention
  Other Names: No intervention

SUMMARY:
Twin pregnancy increases the risk of maternal and fetal complications, which include gestational hypertension, premature labor, twin-to-twin transfusion syndrome, intrauterine growth restriction, anemia, amniotic fluid abnormalities. Comprehensively understanding the molecular mechanisms of the disease and identification of markers contribute to development of novel therapeutic approaches. In addition, the twin pregnancy, especially the monochorionic, is an essential model of "experiments of nature". This model can be applied to distinguish the epigenetic differences of twins in utero and after birth in the same genomic context. The aim of the study is to constitute a prospective cohort of twin pregnancies and the offspring.

DETAILED DESCRIPTION:
Data are collected regarding the pregnancy data of the mother, and mental, physical and sociodemographic information of the offspring. The periods span from diagnosis of twins to 3 years old of the offspring. Biological samples would be collected including maternal blood, placental tissues, cord blood, urine, and stool from the pregnant women or the offspring at the specific time.

The total estimated duration of the study is 6 years, of which the first 2.5 years will correspond to the recruitment period of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age >18 years old.
2. Twin pregnancy.

Exclusion Criteria:

1. Fetal chromosomal or congenital abnormalities.
2. Stillbirth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman with twin pregnancy and their male or female offspring.
Study Population: Woman with twin pregnancy and their offspring within 3 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of maternal and fetal complications | From confirmation of pregnancy to 42 days postpartum
  The incidence of preeclampsia, gestational diabetes mellitus, premature delivery, postpartum hemorrhage, twin to twin transfusion syndrome, selective intrauterine growth restriction.
RNA profiles in placentas of twin pregnancy measured by RNA-sequencing | Immediately after delivery
  Levels of placental RNA expression.
Global DNA methylation in placentas of twin pregnancy measured by whole-genome bisulfite sequencing | Immediately after delivery
  Global DNA methylation levels in placentas of twin pregnancy.
Protein profiles in placentas of twin pregnancy measured by tandem mass tags quantification. | Immediately after delivery
  Levels of proteins in placentas of twin pregnancy.
Post-translation modification of proteins in placentas of twin pregnancy measured by Integrative use of phosphoproteomics, ubiquitylproteomics and acetylproteomics. | Immediately after delivery
  Post-translational levels of proteins in placentas of twin pregnancy.
Metabolite profiles in placentas of twin pregnancy measured by metabolomics | Immediately after delivery
  Metabolite profiles in placentas of twin pregnancy.
Lipid profiles in placentas of twin pregnancy measured by lipidomic analysis | Immediately after delivery
  Lipid profiles in placentas of twin pregnancy.
Predictive protein markers of maternal and fetal complications in maternal blood measured by tandem mass tags quantification | From confirmation of pregnancy to 42 days postpartum
  Levels of specific proteins in maternal blood.
Predictive RNA markers of maternal and fetal complications in maternal blood measured by RNA-sequencing | From confirmation of pregnancy to 42 days postpartum
  Levels of specific RNAs in maternal blood.
Predictive metabolite markers of maternal and fetal complications in maternal blood measured by metabolomics | From confirmation of pregnancy to 42 days postpartum
  Levels of specific metabolites in maternal blood.
Predictive lipid markers of maternal and fetal complications in maternal blood measured by lipidomic analysis | From confirmation of pregnancy to 42 days postpartum
  Levels of specific lipids in maternal blood.

SECONDARY OUTCOMES:
The level of twin Neurodevelopment assessed by Gesell Developmental Schedules | Age at 3 years of the offspring
  The parameters in Gesell Developmental Schedules including adaptive, gross motor, fine motor, language, and social function.
The incidence of long term maternal complications | Three years after delivery
  Including hypertension, diabetes mellitus and metabolic disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No